CLINICAL TRIAL: NCT05545215
Title: Prospective Real-World Clinical Investigation on Dexyane Med® in Adults With Chronic Hand Eczema
Acronym: CARING
Status: Withdrawn | Type: Observational
Why Stopped: no recruitment afetre several months, Sponsor decision
Sponsor: Pierre Fabre Medicament (Industry)
Collaborators: ClinSearch (Other)
Responsible Party: Sponsor
Other Study IDs: NIS12940
Record Dates: First submitted 2022-09-14; First posted 2022-09-19 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2022-08

CONDITIONS: Chronic Hand Eczema

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Dexyane Med: Dexyane MeD® is a non-sterile topical cream, for external use only, available in 30 mL or 100 mL tubes (also available in sample model 5mL tubes).
  Interventions: Device: Dexyane Med

INTERVENTIONS:
Device: Dexyane Med — Dexyane MeD® is a non-sterile topical cream, for external use only, available in 30 mL or 100 mL tubes (also available in sample model 5mL tubes).

SUMMARY:
Prospective, descriptive, multicenter, real-world, international clinical investigation. Data collection is based on current clinical practice over a 6-month follow-up period using both electronic Case Report Form (eCRF) and electronic patient diary (specifically designed mobile/Web application). Based on current clinical practice, at least two milestone visits are anticipated with the possibility of intermediary visits in case of flare recurrence:

* inclusion visit (in-person visit) = Baseline = once clear or almost clear of HE after a moderate to severe flare requiring treatment;
* flare visit(s) (in-person or teleconsultation) = potential intermediary visit(s) required by the patient in case of HE flare, anticipated to occur anytime between inclusion visit and end of study visit;
* end of study visit (in-person or teleconsultation) = regular bi-annual visit for patients' follow-up as per clinical practice, anticipated to occur 6 months post-inclusion (-3 / + 1 months).

DETAILED DESCRIPTION:
This clinical investigation will be a real-world, post-market, prospective, descriptive, multicenter, and international.

The clinical investigation is expected to take place in European countries (France, Spain, Italy, Portugal, and Germany are currently planned). Approximately 200 adult patients from approximately 35 centers (dermatologist practices) will be enrolled and followed for a total duration of 6 months (-3/+1 month). The aim of the study is to describe the patient's practice of Dexyane MeD® in CHE patients, for whom it has been prescribed either alone or in association with Dexyane insulating barrier cream, with no intention of group comparison.

All consecutive patients with moderate to severe CHE who are clear or almost clear of HE after being treated with topical or systemic treatment and who have been prescribed Dexyane MeD® (alone or in association with Dexyane insulating barrier), will be eligible to participate. The study will not provide or recommend any specific treatment procedures; all decisions regarding treatment of included patients will be made by the treating physician in accordance with their usual clinical practice.

Patients' data will be collected by the investigator from the date of prescription of Dexyane MeD® until the end of the observation period (6 months). All patients will be treated and monitored according to the local clinical practice. Based on a feasibility survey among dermatologists in public and/or private practice, at least two milestone visits are anticipated with the possibility of intermediary visits in case of flare recurrence:

* inclusion visit (in-person visit) = Baseline = once clear or almost clear of HE after a moderate to severe flare requiring treatment;
* flare visit(s) (in-person or teleconsultation) = potential intermediary visit(s) required by the patient in case of HE flare, anticipated to occur anytime between inclusion visit and end of study visit;
* end of study visit (in-person or teleconsultation) = regular bi-annual visit for patients' follow-up as per clinical practice, anticipated to occur 6 months post-inclusion (-3 / + 1 months).

Moreover, patients will be provided with all the adequate instructions to complete an electronic patient diary at inclusion (mobile app) and they will be encouraged to complete it throughout the 6-month observation period. Within this digital tool, an additional feature will allow the patient to send pictures of their hands to their physician in case of flare to assess the severity or for the physician to assess response to treatment. The patient will be adequately instructed to focus the picture on the hands only, in order that the picture remain anonymous and no personal data can be collected. The exchange of pictures is a current clinical practice to tackle the lack of appointment availability and has increased exponentially in the last years, in parallel to the increase of remote consultations.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥ 18 years at inclusion.
* Patients diagnosed with CHE (all types of HE admitted: contact, irritative, atopic, etc.) as defined as an eczematous process that lasts for more than three months, or relapses twice or more often per year.
* Patients clear or almost clear of HE at the time of inclusion (i.e., equivalent to a grade 0 or 1 of the IGA scale) after completing treatment (oral or systemic) for a HE flare within the month prior to inclusion.
* Patients having been prescribed with Dexyane MeD® alone or in association with Dexyane insulating barrier cream (the patient can either be a primo-user or a regular user of Dexyane MeD®).
* Patients having provided a signed informed consent.

Exclusion Criteria:

* Patients with another ongoing and evolutive hand skin condition (including psoriasis, and vitiligo).
* Patient with ongoing systemic immunosuppressive therapy.
* Patients participating in interventional trials on any investigational drug at the time of inclusion.
* Patients unable to understand and to comply with the study-related requirements (patient diary to be completed autonomously).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with an initial diagnosis of CHE and having been treated for a moderate to severe flare (i.e., equivalent to a grade 3 or 4 of the IGA scale) and who are clear or almost clear of HE (i.e., equivalent to a grade 0 or 1 of the IGA scale) at the moment of inclusion after treatment by topical or systemic treatment will be eligible for enrollment in the study.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2022-09-07 (Actual); Primary Completion 2022-12-07 (Actual); Study Completion 2022-12-07 (Actual)

PRIMARY OUTCOMES:
Number of days to first relapse of HE after being clear or almost clear of hand eczema | 6 months
  * severity score, and evolution from baseline, of each HE relapse event during the 6-month follow-up using the Investigator Global Assessment (IGA) scale, the modified Total Lesion Symptom Score (mTLSS) and the Chronic Itch Burden Scale
  * number of relapse events observed per patient during the 6-month follow-up;
  * number of days between subsequent HE relapse events during the 6-month follow-up;
  * rate of patients in whom a relapse of HE was observed during the 6-month follow-up.

SECONDARY OUTCOMES:
Description of demographics and clinical profile of included patients | 6 months
  Description of demographics and clinical profile of included patients
Description of scores from the Dermatology Life Quality Index (DLQI) at inclusion and at the end of the 6-month follow-up period. | 6 months
  Description of scores from the Dermatology Life Quality Index (DLQI) at inclusion and at the end of the 6-month follow-up period.
Proportion of patients satisfied with Dexyane MeD® used with or without Dexyane insulating barrier cream, assessed via a specifically adapted questionnaire | 6 months
  Proportion of patients satisfied with Dexyane MeD® used with or without Dexyane insulating barrier cream, assessed via a specifically adapted questionnaire
Proportion of patients adhering to the instructions for use | 6 months
  Proportion of patients adhering to the instructions for use (applications twice a day) on more that 75% of the days for which data are collected. This secondary outcome will be completed by detailed description of variables included in the patient diary and assessing the use of Dexyane MeD® with or without Dexyane insulating barrier cream.
Proportion of patients in whom at least one relevant Adverse Device Effect (ADE) is observed. Relevant ADEs are defined as those leading to Dexyane MeD® or Dexyane insulating barrier cream discontinuation; | 6 months
  Proportion of patients in whom at least one relevant Adverse Device Effect (ADE) is observed. Relevant ADEs are defined as those leading to Dexyane MeD® or Dexyane insulating barrier cream discontinuation;
Description of healthcare resources use due to CHE (consultations and treatment) and impact of CHE on work productivity assessed with the Work Productivity and Activity Impairment (WPAI) questionnaire. | 6 months
  Description of healthcare resources use due to CHE (consultations and treatment) and impact of CHE on work productivity assessed with the Work Productivity and Activity Impairment (WPAI) questionnaire.

IPD SHARING:
Plan to Share IPD: No